CLINICAL TRIAL: NCT05032612
Title: Effects of Photobiomodulation on Postoperative Pain After Primary Endodontic Therapy in Molars With Symptomatic Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Timothy Kirkpatrick, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-DB-21-0579
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pain
Keywords: endodontic treatment; mandibular molar teeth; apical periodontitis.
MeSH Terms: conditions — Pain, Postoperative; Periapical Periodontitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PBM Therapy (Experimental)
  Interventions: Device: PBM Therapy
- PBM Sham (Sham Comparator)
  Interventions: Device: PBM Sham

INTERVENTIONS:
Device: PBM Therapy — After the endodontic treatment, PBM therapy will be performed using a 660 nm diode laser (SiroLaser Advance Plus, Dentsply Sirona Inc, Charlotte, NC, USA), with an 8mm tip diameter.The laser tip will be placed on the following external surfaces in a contact mode: mesiobuccal, distobuccal, mesiolingual and distolingual . The power output of the laser will be 50mW and will be verified by Power Meter (PM600 Power/Energy meter, Molectron Detector Inc, Portland, OR, USA). Each site will be irradiated for 25 s with an energy density of 10 J/cm2 .
  Arms: PBM Therapy
Device: PBM Sham — For the PBM sham similar procedure as PBM therapy will be performed without activating the laser.
  Arms: PBM Sham

SUMMARY:
The purpose of this study is to evaluate the effects of photobiomodulation (PBM) on postoperative pain after endodontic treatment in mandibular molar teeth diagnosed with symptomatic apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Posterior mandibular molars
* No previous root canal therapy on the tooth in question
* Able to complete the endodontic treatment in one visit

Exclusion Criteria:

* Maxillary teeth, mandibular anteriors and premolars
* Infection (swelling, sinus tract) on the tooth in question
* Periodontal disease on the tooth in question
* Dental trauma
* Crown/ root fractures
* Systemic diseases
* Immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryne Jackson, DMD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PBM Therapy | PBM Sham
Started | 17 | 15
Completed | 17 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PBM Therapy | PBM Sham | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.05 (12.83) | 37.7 (14.6) | 41.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 6 | 3 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Pain as Assessed by the Visual Analog Scale
Description: This scale ranges form 0(no pain) to 10(worst pain)
Time Frame: 72 hours after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PBM Therapy | PBM Sham
Number analyzed (Participants) | 17 | 15
score on a scale | 0 (0) | .33 (.48)

2. Secondary Outcome: Pain as Assessed by the Visual Analog Scale
Description: This scale ranges form 0(no pain) to 10(worst pain)
Time Frame: 0 hours, 6 hours, 12 hours and 24 hours hours after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PBM Therapy | PBM Sham
Number analyzed (Participants) | 17 | 15
score on a scale
  0 hours after treatment | 3.94 (2.01) | 6.13 (2.5)
  6 hours after treatment | 1.94 (2.46) | 3.86 (2.7)
  12 hours after treatment | 0.76 (0.90) | 3.33 (2.4)
  24 hours after treatment | 0.23 (0.43) | 1.4 (1.18)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | PBM Therapy | PBM Sham
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT05032612/Prot_SAP_000.pdf